CLINICAL TRIAL: NCT06891248
Title: The Utility of Osteopathic Manipulative Medicine in Weaning Patients from the Ventilator
Brief Title: The Utility of Osteopathic Manipulative Medicine in Weaning Patients from the Ventilator Pilot Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Leslie Ching, Clinical Associate Professor, Oklahoma State University Center for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024193
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Failure; Osteopathy in Diseases Classified Elsewhere
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Subjects in these arms only receive conventional care
- Osteopathic Manipulative Treatment (Experimental): The standard OMM treatment arm includes a 10-minute treatment time for 5 body regions with up to 3 providers working on the patient simultaneously. The OMM attending physician will be physically present and supervising the treatment, and may be participating in the treatment. The 5 body regions include Head, Neck, Thoracic, Ribs, and Abdominal/Diaphragm. The standard technique for the OMM arm includes OA decompression, screening and treating any cervical dysfunction, thoracic inlet myofascial release, rib raising, thoracic paraspinal inhibition, and abdominal diaphragm myofascial release.
  There is an opportunity for an additional 5 minutes of treatment time and additional regions if the lead physician determines it is appropriate based on clinical judgment. The additional 4 regions include Upper Extremity, Lower Extremity, Lumbar, Pelvis, and Sacrum.
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — See treatment arm
  Arms: Osteopathic Manipulative Treatment

SUMMARY:
The objectives of this research are to determine the treatment effect size of OMM to wean patients off of the ventilator, determine the number of patients needed for a larger study (power), determine the willingness of patients/POAs to be recruited, identify the correct dosing of OMM and whether there are concerns for the safety of treatment, and determine whether the hypothesis is feasible for a larger study. The primary outcome measure is the duration of time until a subject is weaned off of mechanical ventilation using Osteopathic Manipulative Medicine (OMM). The secondary outcome measures (see the next section for further explanation) are to determine if OMM affects changes in morbidity and mortality, such as VBG/ABG, NIF, RSBI, P 0.1, FiO2, PEEP, mental status, hemodynamic stability (blood pressure), spontaneous TV, reintubation after extubation, and death.

ELIGIBILITY:
Inclusion Criteria:

1. Acute respiratory failure (hypoxic, hypercapnic, or neuromuscular)
2. Not making satisfactory progress with weaning after being on the ventilator for more than 48 hours
3. Clinical stability for pressure support trial with ventilator to monitor ventilation progression
4. Pulmonology must be following the patient for standardized ventilator management approach and interventions as needed
5. Medical power of attorney (POA) or legally authorized representative (LAR) who is able to consent subject for trial enrollment and treatment
6. Patients who were not referred to the OMM service

Exclusion Criteria:

1. Age less than 18 years old or more than 85 years old
2. BMI>60
3. Moderate/severe neurological disease with expectation of non-progression off the ventilator or poor quality of life predicted (including end-stage dementia with the expectation of non-progression off ventilator, multiple sclerosis, ALS, anoxic brain injury, etc)
4. Status epilepticus or EEG result pending
5. Post-arrest hypothermia protocol
6. Acute stroke
7. Acute rib fractures preventing the implementation of the treatment protocol
8. Acute spinal injury preventing the implementation of the treatment protocol
9. Recent head injury requiring close clinical monitoring
10. Ejection Fraction less than 15%
11. Pleural effusion requiring procedural intervention or inhibiting ventilator progress
12. Pericardial effusion or tamponade requiring procedural intervention or inhibiting ventilator progress
13. ACLS/cardiac arrest within the past 72 hours
14. Confirmed opioid overdose with positive urine drug screen and response to naloxone
15. Patients who were referred to the OMM service

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-06-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Time on ventilator | 90 days
  Number of days that the patient is on the ventilator after inclusion in the study

SECONDARY OUTCOMES:
Ventilator associated measurement | 90 days
  VBG/ABG
Ventilator associated measurement | 90 days
  Negative inspiratory force (NIF)
Ventilator associated measurement | 90 days
  Rapid Shallow Breathing Index (RSBI)
Ventilator associated measurement | 90 days
  Airway occlusion pressure (P0.1)
Ventilator associated measurement | 90 days
  Fraction of inspired oxygen (FiO2)
Ventilator associated measurement | 90 days
  Positive end-expiratory pressure (PEEP)
Blood pressure | 90 days
  Blood pressure
Ventilator associated measurement | 90 days
  Spontaneous Tidal Volume (Spontaneous TV)
Mental status | 90 days
  Whether awake and oriented x 3
Reintubation | 90 days
  Reintubation after extubation
Mortality | 90 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Amber Hood, DFS, Study Director — OSU CHS

IPD SHARING:
Plan to Share IPD: No